CLINICAL TRIAL: NCT03623828
Title: Treating Severe Brain-injured Patients With Apomorphine: a Behavioral and Neuroimaging Study
Brief Title: Treating Severe Brain-injured Patients With Apomorphine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Liege (Other)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Steven Laureys, Principal Investigator, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/81a
Record Dates: First submitted 2018-07-25; First posted 2018-08-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Disorder of Consciousness
Keywords: unresponsive wakefulness syndrome; minimally conscious state; apomorphine; crs-r
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State | interventions — Apomorphine

STUDY DESIGN:
Intervention Model Description: This is an open-label single-arm prospective pilot study. Included patients all undergo the same study protocol.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apomorphine treatment (Experimental): Treatment by apomorphine hydrochloride subcutaneous infusion 12 hours per day during 30 days: 5-days titration phase (increasing doses from 0 to 4 mg/h), 7 days of maintenance at 4 mg/h and 18 days of maintenance phase with possible increase up to 6 mg/h if well tolerated.
  Two days before the initiation of apomorphine, domperidone 20mg t.i.d per os (or via gastric tube) will be initiated to reduce common side effects. It will be maintained at least 7 days before an optional tapering off in the absence of nausea of vomiting.
  Interventions: Drug: Apomorphine Hydrochloride 50Mg/10mL Prefilled Syringe

INTERVENTIONS:
Drug: Apomorphine Hydrochloride 50Mg/10mL Prefilled Syringe — Product administered using an external continuous subcutaneous infusion pump.
  Other Names: APO-go PFS 5mg/ml

SUMMARY:
Background:

Patients who survive severe brain injury may develop chronic disorders of consciousness. Treating these patients to improve recovery is extremely challenging because of scarce and inefficient therapeutical options.

Among pharmacological treatments, apomorphine, a potent direct dopamine agonist, has exhibited promising behavioral effects, but its true efficacy and its mechanism remains unknown. This pilot study aims to verify the effects of apomorphine subcutaneous infusion in patients with disorders of consciousness, investigate the neural networks targeted by this treatment and evaluate the feasibility of a larger double-blind randomized placebo-controlled trial.

Methods/design:

This study is a prospective open-label pilot clinical trial. Six patients diagnosed with disorders of consciousness will be included to receive a 4-weeks regimen of daily subcutaneous infusions of apomorphine hydrochloride. Patients will be monitored for four weeks before the initiation of the therapy, closely during treatment and they will undergo a 4-weeks inpatient follow-up after washout, as well as a two-year long-term remote follow-up. Shortly before and after the treatment regimen, the subjects will receive a multimodal assessment battery including neuroimaging exams.

Primary outcome will be determined as behavioral response to treatment as measured by changes of diagnosis using the Coma Recovery Scale - Revised (CRS-R), while secondary outcome measures will include the Nociception Coma Scale - Revised (NCS-R, circadian rhythm modifications using actimetry, core body temperature recording and night electroencephalography (EEG), positron emission tomography (PET), resting-state high-density EEG and functional magnetic resonance imaging (fMRI). The Glasgow Outcome Scale - Extended (GOS-E) and a phone-adapted version of the CRS-R will be used for long-term follow-up.

Statistical analyses will focus on the detection of changes induced by apomorphine treatment at the individual level (comparing data before and after treatment) and at the group level (comparing responders with non-responders). Response to treatment will be measured at four different levels: 1. behavioral response (CRS-R, NCS-E, GOS-E), 2. brain metabolism (PET), 3. network connectivity (resting-state fMRI and high-density EEG) and 4. Circadian rhythm changes (actimetry, body temperature, night EEG).

Discussion:

Apomorphine is a promising and safe candidate for the treatment of disorders of consciousness but its efficacy, the profile of the responding population and its underlying mechanism remain to be determined. This pilot study will provide unprecedented data that will allow to investigate the response to apomorphine using multimodal methods and shed new light on the brain networks targeted by this drug in terms of metabolism, functional connectivity and behavioral response. The investigators aim to better define the phenotype of potential responders to identify them more easily and develop personalized patient management. This preliminary study will lay ground for a subsequent larger-scale placebo-controlled double-blind trial which will provide quantitative data on effect size controlled for spontaneous recovery.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old.
* Clinically stable, not dependent on medical ventilators for respiration.
* Diagnosed as in an unresponsive wakefulness syndrome or minimally conscious state according to the international criteria and based on at least 2 consistent CRS-R in the last 14 days (one CRS-R in the last 7 days).
* More than 6 weeks post-insult (starting the apomorphine treatment at 10 weeks minimum)
* No serious neurological impairments others than related to their acquired brain injury.
* No neurological medications other than anti-epileptic or anti-spasticity drugs within the last two weeks.
* No use of dopaminergic medications other than apomorphine within the last two weeks.
* Informed consent from legal representative of the patient (if patients recover, their consent will also be obtained).

Exclusion Criteria:

* Use of dopamine agonists or antagonists (e.g. amantadine, bromocriptine, l-dopa, pramipexole, ropinirole, amphetamine, bupropion, methylphenidate / risperidone, haloperidol, chlorpromazine, flupentixol, clozapine, olanzapine, quetiapine) in the last 4 weeks or 4 half-lives of the drug.
* Use of drugs with known significant prolongation of the QT interval (e.g. class 1 antiarrythmics, sotalol, macrolides, quinolones, antipsychotic drugs, tricyclic antidepressants. Methadone, chloroquine, quinine)
* A corrected QT interval over 480ms (calculated using Bazett's formula on a standard 12-lead ECG recorded in the last 14 days) or other risk factors for arrhythmia (congestive cardiac failure, severe hepatic impairment or significant electrolyte disturbance).
* A history of previous neurological functional impairment.
* Contraindication to MRI, EEG, or PET (e.g., electronic implanted devices, active epilepsy, external ventricular drain).
* Use of nitrates or other vasodilators, central nervous system acting agents such as barbiturates, morphine and related drugs (relative exclusion criterion)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2022-11-13 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Coma Recovery Scale - Revised (CRS-R) | up to 90 days (10x before treatment, 6x during treatment and 5x after treatment)
  The CRS-R is a standardized validated neurobehavioral scale designed to assess patients with disorders of consciousness. It is divided in 6 subscales: Auditory Function (0-4 points), Visual Function (0-5 points), Motor Function (0-6 points), Oromotor/Verbal Function (0-3 points), Communication (0-2 points), Arousal (0-3 points). The subscores are summed to calculate a total score ranging from 0 to 23 points. Higher scores indicate better functions. More importantly, it provides the patient's diagnosis (coma, UWS, MCS-, MCS+, EMCS) based on the presence of specific items in different subscales (regardless of total score). Analyses will look for changes of diagnosis, changes of total score and changes of each subscore before, during and after apomorphine treatment.

SECONDARY OUTCOMES:
Nociception Coma Scale - Revised (NCS-R) | up to 90 days (5x before treatment, 4x during treatment and 5x after treatment)
  The NCS-R is a standardized validated scale designed to assess the perception of pain in patients with disorders of consciousness unable to functionally communicate. It is divided in 3 subscales: Motor Response (0-3 points), Verbal Response (0-3 points) and Facial Expression (0-3 points). The subscores are summed to calculate a total score ranging from 0 to 9 points. Higher scores indicate a higher perception of pain. Analyses will look for changes of total score and changes of each subscore before, during and after apomorphine treatment.
resting-state EEG | up to 90 days (4x before treatment, 4x during treatment and 4x after treatment)
  Changes in EEG spectral power within fixed bands or dynamic connectivity using median spectral connectivity and graph-theoretic topology metrics (clustering coefficient, path length, modularity and participation coefficient) after apomorphine treatment.
EEG with auditory paradigms | up to 90 days
  Multivariate classifier giving the probabilty to have signs of consciousness based on a machine-learning approach using 120 EEG markers.
PET | up to 90 days (1x before treatment and 1x after treatment)
  Changes in quantification of PET signal using standardized uptake values of fluorodeoxyglucose after apomorphine treatment.
fMRI | up to 90 days (1x before treatment and 1x after treatment)
  Changes in MRI functional connectivity using a seed-voxel approach, between regions of interest (here: striatum, globus pallidus interna, thalamus and prefrontal cortex) and the time course from all other brain voxels, after apormorphine treatment
Circadian rythmycity using body movements | constant recording from enrollment up to 90 days
  We use wrist actigraph recorded data on limb movements to calculate circadian rythmycity, measured in minutes. It corresponds to the period of the biological temporal rhythms with oscillations around 24 hours.
Circadian rythmycity using body temperature variations | constant recording from enrollment up to 90 days
  We use data recorded from non-invasive body temperature measurement devices to calculate circadian rythmycity, measured in minutes. It corresponds to the period of the biological temporal rhythms with oscillations around 24 hours.
Number of sleep cycles using night EEG | actimetry and core body temperature recorded during the whole study; night EEG 1x before treatment initiation and 1x after treatment withdrawal
  We use data measured with whole-night EEG recordings to calculate the number of sleep cycles during one night and the duration spent in each phase of sleep.
Glasgow Outcome Scale - Extended (GOS-E) | from 6 months post-treatment up to 24 months post-treatment (1x at 6 months, 1x at 12 months, 1x at 24 months)
  The GOS-E is a standardized validated scale designed to assess the the functional outcome of patients with disorders of consciousness. It is a single score ranging from 1 (dead) to 8 (upper good recovery). Higher scores indicate a higher functional recovery. It will be performed remotely by telephone contact with the patient or their relatives.
  Analyses will look at differences in GOS-E score between responders and non-responders to apomorphine treatment, as well as differences in time within individual patients.
Phone-adapted CRS-R | from 6 months post-treatment up to 24 months post-treatment (1x at 6 months, 1x at 12 months, 1x at 24 months)
  The phone-adapted CRS-R is a scale designed to assess remotely patients with disorders of consciousness. Unlike the CRS-R, it does not comprise subcores or a total score, but provides the clinical diagnosis of the patient (coma, UWS, MCS-, MCS+, EMCS) using the same diagnostic items as the CRS-R.
  Analyses will look at differences in Phone-adapted CRS-R diagnosis between responders and non-responders to apomorphine treatment, as well as differences in time within individual patients.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Laureys, M.D., Ph.D., Principal Investigator — University hospital of Liège
Locations (2):
- Belgium (2):
  - Neurological Hospital Center William Lennox, Ottignies, Brabant Wallon
  - University Hospital of Liège, Liège

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fridman EA, Calvar J, Bonetto M, Gamzu E, Krimchansky BZ, Meli F, Leiguarda RC, Zafonte R. Fast awakening from minimally conscious state with apomorphine. Brain Inj. 2009 Feb;23(2):172-7. doi: 10.1080/02699050802649662. PMID 19191097
- [Background] Fridman EA, Krimchansky BZ, Bonetto M, Galperin T, Gamzu ER, Leiguarda RC, Zafonte R. Continuous subcutaneous apomorphine for severe disorders of consciousness after traumatic brain injury. Brain Inj. 2010;24(4):636-41. doi: 10.3109/02699051003610433. PMID 20235766
- [Background] Gosseries O, Charland-Verville V, Thonnard M, Bodart O, Laureys S, Demertzi A. Amantadine, apomorphine and zolpidem in the treatment of disorders of consciousness. Curr Pharm Des. 2014;20(26):4167-84. PMID 24025057
- [Derived] Sanz LRD, Lejeune N, Szymkowicz E, Bonin EAC, Panda R, Sala A, Thibaut A, Huerta-Gutierrez R, Dardenne N, Dikenstein D, Van Goethem S, Ledoux D, Hustinx R, Stender J, Farber NM, Zafonte RD, Schiff ND, Laureys S, Gosseries O. Apomorphine for prolonged disorders of consciousness: a multimodal open-label study. EClinicalMedicine. 2024 Nov 15;78:102925. doi: 10.1016/j.eclinm.2024.102925. eCollection 2024 Dec. PMID 39624459
- [Derived] Sanz LRD, Lejeune N, Blandiaux S, Bonin E, Thibaut A, Stender J, Farber NM, Zafonte RD, Schiff ND, Laureys S, Gosseries O. Treating Disorders of Consciousness With Apomorphine: Protocol for a Double-Blind Randomized Controlled Trial Using Multimodal Assessments. Front Neurol. 2019 Mar 19;10:248. doi: 10.3389/fneur.2019.00248. eCollection 2019. PMID 30941094